CLINICAL TRIAL: NCT03505138
Title: Impact of Telemedicine in the Rate of Readmission for COPD and Cost-effectiveness Analysis (e- Pneumo ) : Project CRONEX 3.0
Brief Title: Impact of Telemedicine in the Rate of Readmission for COPD. Project CRONEX 3.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Jaime Corral Penafiel, Medical Doctor, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CRONEX3.0
Record Dates: First submitted 2018-03-05; First posted 2018-04-23 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2018-04

CONDITIONS: COPD
Keywords: COPD; hospitalization; telemedicine platform
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Delivery of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group intervention (Experimental): Conventional management for COPD will take place in our health care system more telematics intervention.
  Interventions: Device: Group intervention
- Group control (Active Comparator): Is performed only conventional management of COPD in our health care system.
  Interventions: Other: health care system

INTERVENTIONS:
Device: Group intervention — GROUP 1 (telematic group):
  These patients will have a tablet connected via internet (Telefónica-e-Health). They have to measure their lung function, temperature, pulse oxymetry and symtoms questionnaire every week. The device (tablet) asks them about possible COPD exacerbation. If the patient has an exacerbation, the device offers them a treatment for this exacerbation and it begins a following of this exacerbation until resolution, every day.
  The pneumologists will receive an alert in other tablet when the patients have an exacerbation or worsening of their diseases.
  The period of monitoring is 1 year.
  Other Names: Telematic intervention
  Arms: Group intervention
Other: health care system — GROUP 2 (conventional group or control group) Patients with a COPD exacerbation can go to their family physicians or emergency services and these physicians will establish a treatment and a monitoring of these exacerbation (conventional group).
  The period of monitoring is 1 year.
  Arms: Group control

SUMMARY:
The prevalence of COPD is high and suppose one of the first public health problem in the world. It has a high morbidity and mortality and healthcare costs. The economic aspect is directly related to hospitalization, accounting for 45-50% of total expenditure of COPD. Patients with frequent exacerbations generate most of the cost.

In these patients, there are not standardized treatments or monitoring in a medium or long term, but it seems reasonable that the combination of various interventions (programs self-care, active role of health professionals in consultations, home programs, group visits, establishment action plans for patients, use of communication technologies or social networks) may improve many patient outcomes.

The hypothesis of our work will be to introduce telemedicine platform to establish action plans for the patient, recognition of symptoms and exacerbations, treatments for the exacerbations, training material on COPD, smoking and inhalation therapy, establishment of a fast and fluid communication with pulmonologist, with the purpose of responding to various health problems that patients with COPD (exacerbator phenotype or ACO phenotype) may have. We will study the impact of this tool to reduce the rate income or readmission for the patients with COPD, analyzing it from the perspective of cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. COPD, which after evaluation of its clinical history, belonging to exacerbator phenotype (chronic bronchitic / emphysema) or mixed phenotype ("COPD-asthma") readmission (2 or more income in the previous year) and are stable least six weeks before inclusion in the study.
2. Age over 18 years
3. The patient or caregiver should be able to use the tablet type telematic tool for tracking and monitoring.

Exclusion Criteria:

1. Patients with severe comorbidity grade IV heart failure, renal failure on hemodialysis or active neoplasia
2. Patients with difficulties phone coverage
3. Patients with lack of adequate social and family support.
4. Patients who do not grant informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Assess whether a telematic program intervention can decrease the rate of readmissions in patients with COPD, comparing with conventional management. | one year
  outcome measure: the rate of readmissions during the study

SECONDARY OUTCOMES:
Conducting a cost-effectiveness study that allows us to estimate the incremental cost-effectiveness ratio (ICER) of this patient group compared with the control group. | one year
  outcome measure: incremental cost-effectiveness ratio (ICER) between these two arms
Compare the quality of life of COPD patients by measuring CAT in study groups | one year
  outcome measure: quality of life measured by CAT questionnaire
To study the evolution of lung function in both groups after 1 year of follow up. | one year
  outcome measure: lung function by spirometry (FEV1/FVC, FVC, FEV1)
Analyze the survival at 12 months follow-up in each group. | one year
  outcome measure: number of deaths in each group to see the survival in this study
Analyze a biomarker predictor of exacerbation severity. | one year
  outcome measure: PCR (mg/L)
Analyze the inhaler compliance and adherence of treatment in both groups. | one year
  outcome measure: Morisky-Green´s scoring
Make satisfaction survey patients and caregivers, comparing both study groups. | one year
  outcome measure: satisfaction (very satisfied, satisfied, unsatisfied, very unsatisfied)
Compare the quality of life of patients by measuring EQ-5D in study groups | one year
  outcome measure: EQ-5D questionnaire
Analyze a biomarker predictor of exacerbation severity. | one year
  outcome measure: fibrinogen (g/L)
Analyze a biomarker predictor of exacerbation severity. | one year
  outcome measure: leukocytes (mil/mm3)
Analyze a biomarker predictor of exacerbation severity. | one year
  outcome measure: eosinophils (mil/mm3)
Analyze a biomarker predictor of exacerbation severity. | one year
  outcome measure: pro-BNP (pg/ml)
Analyze a biomarker predictor of exacerbation severity. | one year
  outcome measure: cholesterol (mg/dL)
Analyze a biomarker predictor of exacerbation severity. | one year
  outcome measure: proteins (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Corral, MD, Principal Investigator — Hospital San Pedro de Alcántara. Cáceres. Spain
Locations (1):
- Jaime Corral Peñafiel, Cáceres, Spain

REFERENCES:
- [Background] Cosio BG, Agusti A. Update in chronic obstructive pulmonary disease 2009. Am J Respir Crit Care Med. 2010 Apr 1;181(7):655-60. doi: 10.1164/rccm.201001-0111UP. No abstract available. PMID 20335383
- [Background] Escarrabill J. Discharge planning and home care for end-stage COPD patients. Eur Respir J. 2009 Aug;34(2):507-12. doi: 10.1183/09031936.00146308. PMID 19648525
- [Background] Hurst JR, Fitzgerald-Khan F, Quint JK, Goldring JJ, Mikelsons C, Dilworth JP, Wedzicha JA. Use and utility of a 24-hour Telephone Support Service for 'high risk' patients with COPD. Prim Care Respir J. 2010 Sep;19(3):260-5. doi: 10.4104/pcrj.2010.00035. PMID 20571731
- [Background] Bourbeau J, Julien M, Maltais F, Rouleau M, Beaupre A, Begin R, Renzi P, Nault D, Borycki E, Schwartzman K, Singh R, Collet JP; Chronic Obstructive Pulmonary Disease axis of the Respiratory Network Fonds de la Recherche en Sante du Quebec. Reduction of hospital utilization in patients with chronic obstructive pulmonary disease: a disease-specific self-management intervention. Arch Intern Med. 2003 Mar 10;163(5):585-91. doi: 10.1001/archinte.163.5.585. PMID 12622605
- [Background] Jurado Gamez B, Feu Collado N, Jurado Garcia JC, Garcia Gil F, Munoz Gomariz E, Jimenez Murillo L, Munoz Cabrera L. Home intervention and predictor variables for rehospitalization in chronic obstructive pulmonary disease exacerbations. Arch Bronconeumol. 2013 Jan;49(1):10-4. doi: 10.1016/j.arbres.2012.08.003. Epub 2012 Oct 22. English, Spanish. PMID 23089685
- [Background] De Vries B, Darling-Fisher C, Thomas AC, Belanger-Shugart EB. Implementation and outcomes of group medical appointments in an outpatient specialty care clinic. J Am Acad Nurse Pract. 2008 Mar;20(3):163-9. doi: 10.1111/j.1745-7599.2007.00300.x. PMID 18336693
- [Background] Bischoff EW, Hamd DH, Sedeno M, Benedetti A, Schermer TR, Bernard S, Maltais F, Bourbeau J. Effects of written action plan adherence on COPD exacerbation recovery. Thorax. 2011 Jan;66(1):26-31. doi: 10.1136/thx.2009.127621. Epub 2010 Oct 30. PMID 21037270